CLINICAL TRIAL: NCT03465579
Title: Multi-cohort Investigational Study to Evaluate the Impact of Pelvic Mp-3TMRI and Whole-body 68Ga-PSMA PET/CT for Diagnosis of Clinically-significant Prostate Cancer and Pre-surgical Staging.
Brief Title: Mp-3TMRI and 68Ga-PSMA PET/CT Guided Prostate Biopsy and Tumor Node Metastasis (TNM) Staging.
Acronym: BIOPSTAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients in cohort 1 continued for prolonged periods given the difficulties encountered in the COVID period and to date in this setting evidence has already developed that reduces the the innovativeness of the project.
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRST185.05
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: 68Ga-PSMA PET/CT Guided Prostate Biopsy; Mp-3TMRI Guided Prostate Biopsy; Prostate Cancer; TNM Staging; Diagnosis
Keywords: Diagnosis Prostate Cancer; TNM staging; 68Ga-PSMA PET/CT guided prostate biopsy; mp-3TMRI guided prostate biopsy; pre-surgical staging; clinically-suspected prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Other): Men with suspected clinically-significant PCa (CS-PCa) who are candidates for prostate biopsy or after first-round negative transrectal ultrasonography (TRUS) biopsy
  Interventions: Diagnostic Test: pelvic MRI; Diagnostic Test: 68Ga-PSMA PET/CT
- Cohort 2 (Other): Men framed in Active Surveillance (PRIAS study), scheduled for PRIAS repeat biopsy.
  Interventions: Diagnostic Test: pelvic MRI; Diagnostic Test: 68Ga-PSMA PET/CT
- Cohort 3a (Other): Men with high-risk PCa (HR-PCa) prior to radical surgery.
  Interventions: Diagnostic Test: pelvic MRI; Diagnostic Test: 68Ga-PSMA PET/CT
- Cohort 3b (Other): Men diagnosed with CS-PCa prior to nerve-sparing prostate surgery (NSS).
  Interventions: Diagnostic Test: pelvic MRI; Diagnostic Test: 68Ga-PSMA PET/CT

INTERVENTIONS:
Diagnostic Test: pelvic MRI — multi-parametric pelvic MRI
Diagnostic Test: 68Ga-PSMA PET/CT — 68Ga-PSMA PET/CT

SUMMARY:
BIOPSTAGE is a prospective, non-randomized, diagnostic, multi-cohort investigational study to evaluate the impact of pelvic Multi-parametric 3-Tesla magnetic resonance imaging (mp-3TMRI) and whole-body 68Ga-PSMA PET/CT for diagnosis of clinically-significant prostate cancer and pre-surgical staging.

DETAILED DESCRIPTION:
The aim of this study is to characterize the diagnostic accuracy of both multi-parametric pelvic Magnetic Resonance Imaging (MRI) (T2-weighted, Diffusion Weighted Imaging (DWI), Dynamic Contrast Enhancement (DCE) and 68Ga-chelated Prostate Specific Membrane Antigen ligand (68Ga-PSMA) Positron Emission Tomography/Computed Tomography (PET /CT) in three cohorts of patients:

* COHORT 1 Guiding prostate biopsies in men with clinical suspicion and/or unconfirmed clinically-significant prostate cancer (CS-PCa) on initial prostate biopsy;
* COHORT 2 Targeting repeat prostate biopsy in patients on Active Surveillance (PRIAS Study), scheduled for PRIAS repeat biopsy;
* COHORT 3

Providing pelvic / whole-body pre-surgical staging in:

* 3a: men with high-risk PCa (HR-PCa);
* 3b: men candidates for nerve sparing surgery (NSS);

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 - Biopsy guidance in clinically-suspected PCa

1. Men aged 45 to 75 years old with clinically-suspected PCa candidated for either initial or repeat TRUS-guided prostate biopsy, meeting any of the following criteria:

a) Abnormal PSA metrics, defined as follows:

A rising and/or persistently elevated serum PSA (i.e PSA > 2.5ng/ml for men in the age group comprising 60 to 75 years old; PSA > 3.0ng/ml for men in the age group comprising 45 to 60 years old) and at least one of the following PSA-based metrics:

i. Percent free PSA (%fPSA) < 25% with PSA range 4-10ng/ml (NCCN); ii. PSA velocity (PSAvel) >0.35 ng/mL/y; iii. PSA density (PSAden) > 0.25ng/mL/cc iv. PSA > 10ng/ml, 50% risk of PCa (EAU) b) Suspicious digital rectal examination (DRE), 5-30% risk of PCa; c) Prostate Cancer Gene 3 (PCA3) > 35; d) Suspicious findings on first-round biopsy: i. A few Atypical Glands immediately adjacent to HG-PIN, 50% risk of PCa; ii. Atypical Small Acinar Proliferation, 40% of PCa; iii. Multifocal High-Grade Prostatic intraepithelial neoplasia (HG-PIN), 30% ; iv. Intraductal carcinoma as solitary finding, 90% of PCa;

Cohort 2 - Biopsy guidance on Active Surveillance

Men consenting to enter the PRIAS MRI side-study as per currently inclusion criteria in Version Number 1.0 dated August 20, 2013. These are:

1. Histologically-proven adenocarcinoma of the prostate;
2. Age ≥ 18
3. Men should be fit for curative treatment;
4. Clinical stage T1c or T2;
5. Gleason score 3+3=6;
6. One or two biopsy cores invaded with prostate cancer:

   1. If an MRI, including targeted biopsies on positive lesions, is done at inclusion, there is no limit in the number of positive cores (that is, more than two, and no limit in the % of cancer present in the cores);
   2. If saturation biopsies (either trans-perineal or trans-rectal) are done 15% of the cores can be positive with a maximum of 4 (i.e. 26 cores 4 cores can be positive) (all other inclusion criteria still apply);
7. PSA density (PSA D) less than 0.2;
8. PSA-level at diagnosis ≤ 10 ng/mL;

Cohort 3a - Pre-surgical TNM staging in high-risk prostate cancer

1. Male, aged 18 years or older;
2. Cyto / histological confirmation of PCa (i.e. TRUS-guided biopsies; TURP);
3. Any of the PCa high risk features for Organ-Confined Disease (OCD):

   * Clinical T stage ≥ T2c;
   * Gleason Score ≥ 8;
   * Serum PSA > 20 ng/mL;
4. Any of the PCa high-risk features for Locally-Advanced Disease (LAD):

   * Clinical T stage ≥ T3b-T4 OR any T and clinical N1 disease;
   * Gleason Score ≥ 8;
   * Serum PSA > 20 ng/mL;
5. Routine clinical staging (CTscan ± Bone scan) performed within 12 weeks enrolment returning negative or equivocal results for distant metastatic disease;

Cohort 3b - pelvic TNM staging of prostate cancer prior to nerve-sparing radical prostatectomy

1. Male, aged 18 years or older;
2. Cyto / histological confirmation of PCa (i.e. TRUS-guided biopsies; TURP);
3. All of the following PCa-related features must be met for nerve-sparing (either mono- or bi-lateral):

   * Clinical T stage ≤ T2b;
   * Gleason Score ≤ 7 (3+4) and maximum one biopsy with Gleason > 6 at the ipsilateral side;
   * Serum PSA < 10 ng/mL;

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

1. Hormone androgen deprivation therapy of any type within 6 months prior to enrollment.
2. Prior pelvic radiotherapy;
3. Sickle cell disease;
4. Insufficient renal function (eGFR < 30 mL/min/1.73 m2);
5. Hip prosthesis, vascular grafting or other conditions affecting imaging;
6. Contraindication to MRI, including but not restricted to: pacemaker or other electronic im-plants, known metal in the orbit, MR incompatible surgical or cerebral aneurysm clips, shrapnel, tattoos, non-removable body piercings (relative contraindications);
7. History of allergic reactions attributed to compounds of similar chemical or biologic com-position to 68Ga-PSMA or Gadolinium-based contrast agents used in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
sensitivity of both 68Ga-PSMA PET/CT and mp-3TMRI imaging | up to 36 months
  sensitivity of both 68Ga-PSMA PET/CT and mp-3TMRI imaging will be calculated as the ratio between the number of positive cases at 68Ga-PSMA PET/CT or mp-3TMRI and number of patients who underwent to these exams
specificity of both 68Ga-PSMA PET/CT and mp-3TMRI imaging | up to 36 months
  specificity will be calculated considering negative cases at 68Ga-PSMA PET/CT or mp-3TMRI and number of patients who underwent to these exams
Positive predictive value of both 68Ga-PSMA PET/CT and mp-3TMRI imaging | up to 36 months
  Positive predictive value will be calculated considering the ratio between positive patient at 68Ga-PSMA PET/CT/mp-3TMRI confirmed as positive throughout biopsy and overall positive patient at 68Ga-PSMA PET/CT/mp-3TMRI
negative predictive value of both 68Ga-PSMA PET/CT and mp-3TMRI imaging | up to 36 months
  negative predictive value will be calculated considering the ratio between negative patient at 68Ga-PSMA PET/CT/mp-3TMRI confirmed as negative throughout biopsy and overall negative patient at 68Ga-PSMA PET/CT/mp-3TMRI

SECONDARY OUTCOMES:
Incidence of adverse events | up to 30 days following study procedures
  The number and percentage of treated patients undergoing grade 1 to 4 adverse events will be tabulated for each cohort and diagnostic procedure, using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 should be used to assess and grade AE severity.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Matteucci, Study Chair — IRST IRCCS
Locations (2):
- Italy (2):
  - AUSL della Romagna, Forlì, FC
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC